CLINICAL TRIAL: NCT02729753
Title: Clinical Study to Evaluate the CryoBalloon™ Full and Swipe Ablation Systems for Ablation of Human Esophageal Epithelium
Brief Title: Clinical Study to Evaluate CryoBalloon™ Full and Swipe Ablation Systems for Ablation of Human Esophageal Epithelium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP0014
Record Dates: First submitted 2016-03-09; First posted 2016-04-06 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2018-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CryoBalloon™ Full Ablation System (Other): To evaluate CryoBalloon™ Full Ablation System for the ablation of 360 degrees of human esophageal epithelium in patients scheduled to undergo esophagectomy.
  Interventions: Device: CryoBalloon™ Full Ablation System
- CryoBalloon™ Swipe Ablation System (Other): To evaluate CryoBalloon™ Swipe Ablation System for the ablation of 90 degrees of human esophageal epithelium in patients scheduled to undergo esophagectomy.
  Interventions: Device: CryoBalloon™ Swipe Ablation System

INTERVENTIONS:
Device: CryoBalloon™ Full Ablation System — Tissue Ablation using CryoBalloon™ Full Ablation System
  Other Names: CryoBalloon Ablation System (360)
  Arms: CryoBalloon™ Full Ablation System
Device: CryoBalloon™ Swipe Ablation System — Tissue Ablation using CryoBalloon™ Swipe Ablation System
  Other Names: CryoBalloon Ablation System (90)
  Arms: CryoBalloon™ Swipe Ablation System

SUMMARY:
This study will evaluate the C2 CryoBalloon™ Full and Swipe Ablation Systems for the ablation of human esophageal epithelium in patients scheduled to undergo esophagectomy for reasons unrelated to the objective of the study

DETAILED DESCRIPTION:
The primary outcomes for the study are the safety and treatment effect of the C2 CryoBalloon™ Ablation System. An esophagectomy will be performed as scheduled following the ablation procedure; histopathological analysis of surgically-resected specimens will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of one 3cm area of non-ulcerated columnar-lined esophagus or squamous-lined tissue suitable for ablation
* Older than 18 years of age
* Requires a clinically necessary esophagectomy for esophageal cancer or other indications.

Exclusion Criteria:

* Patient has esophageal narrowing limiting access to the intended sites of ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Louie, MD, Principal Investigator — Swedish Medical Center and Cancer Institute
Locations (2):
- United States (2):
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Medical Center and Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for esophagectomy for esophageal cancer or other indications unrelated to the objective of this study were approached to allow for use of cryoballoon ablation in area to be resected prior to surgery.
Groups:
- CryoBalloon Swipe Ablation System: To evaluate CryoBalloon™ Full Ablation System for the ablation of 90 degrees of human esophageal epithelium in patients scheduled to undergo esophagectomy.
Period: Overall Study
Arm/Group | CryoBalloon™ Full Ablation System | CryoBalloon Swipe Ablation System
Started | 3 (First patient enrolled April 2016) | 7 (First patient enrolled April 2016)
Completed | 3 (Study Complete on 30 Oct 2016) | 6 (Study Complete on 30 Oct 2016)
Not Completed | 0 | 1
Not completed — Device Malfunction. No units in stock. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CryoBalloon™ Swipe Ablation System: To evaluate CryoBalloon™ Full Ablation System for the ablation of 90 degrees of human esophageal epithelium in patients scheduled to undergo esophagectomy.
- Total: Total of all reporting groups
Arm/Group | CryoBalloon™ Swipe Ablation System | CryoBalloon™ Full Ablation System | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [58 to 77] | 57 [51.5 to 66] | 64 [58 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 1 | 6
  Netherlands | 1 | 2 | 3
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.3 [22 to 26.9] | 23.3 [20.5 to 24.2] | 26 [23.9 to 26.7]
History of GERD [Count of Participants; unit: Participants] | 4 | 1 | 5
History of Barrett's Esophagus [Count of Participants; unit: Participants] | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety of the CryoBalloon™ Full and Swipe Ablation System
Description: Number of participants with serious, device-related adverse events after treatment with the CryoBalloon™ Swipe Ablation System
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CryoBalloon™ Swipe Ablation System | CryoBalloon™ Full Ablation System
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

2. Primary Outcome: Effect of Ablation to Submucosa at Different Depth of Tissue Ablation Using the CryoBalloon™ Full and Swipe Ablation Systems
Description: Evaluated by depth and uniformity of ablation effect in the esophagus based on histopathologic assessment.
  Dose response by effect of ablation to submucosa:
  0: Normal
  1. Inflammatory cell infiltration
  2. Separation with inflammation
  3. Edema and Necrosis
Time Frame: 2 weeks
Population: Submucosal evaluation done for patients at differing doses.
Measure: Number; unit: units on a scale
Arm/Group | CryoBalloon™ Full Ablation System | CryoBalloon™ Swipe Ablation System
Number analyzed (Participants) | 3 | 6
units on a scale
  0.5mm/sec : Immediate esophagectomy: number analyzed (Participants) | 1 | 1
  0.5mm/sec : Immediate esophagectomy | 2 | 0
  0.5mm/sec : Esophagectomy 5 days Post: number analyzed (Participants) | 1 | 1
  0.5mm/sec : Esophagectomy 5 days Post | 3 | 1
  0.6mm/sec : Immediate esophagectomy: number analyzed (Participants) | 1 | 1
  0.6mm/sec : Immediate esophagectomy | 1 | 2
  0.8mm/sec :Immediate esophagectomy: number analyzed (Participants) | 0 | 1
  0.8mm/sec :Immediate esophagectomy |  | 2
  0.8mm/sec : Esophagectomy 5 days Post: number analyzed (Participants) | 0 | 1
  0.8mm/sec : Esophagectomy 5 days Post |  | 1
  0.9mm/sec : Immediate esophagectomy: number analyzed (Participants) | 0 | 1
  0.9mm/sec : Immediate esophagectomy |  | 1

3. Secondary Outcome: Device Performance: Average Procedure Time
Description: Average Procedure time as measured from start to finish of ablation.
Time Frame: Minutes from start to end of procedure
Measure: Mean (Full Range); unit: Minutes
Arm/Group | CryoBalloon™ Full Ablation System | CryoBalloon™ Swipe Ablation System
Number analyzed (Participants) | 3 | 6
Minutes | 5 [5 to 5] | 4.8 [1 to 10]

4. Secondary Outcome: Device Performance: Ease of Deployment of Device
Description: Likert Scale measuring physician satisfaction. 0 (worst) to 10 (best)
Time Frame: Minutes, from start to end of procedure
Population: CryoBalloon Full and Swipe Ablation Systems used by physicians to perform ablation
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CryoBalloon™ Full Ablation System | CryoBalloon™ Swipe Ablation System
Number analyzed (Participants) | 3 | 6
units on a scale | 9 [9 to 9] | 7.8 [7 to 9]

ADVERSE EVENTS:
Arm/Group | CryoBalloon™ Full Ablation System | CryoBalloon™ Swipe Ablation System
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CryoBalloon™ Full Ablation System (N=3) | CryoBalloon™ Swipe Ablation System (N=6)
Post Procedure Pain (General disorders) | 1 (1) | 0 (0) — Patient experienced pain score of 3 on VAS scale 0 - 10, 24 hours post procedure.

LIMITATIONS AND CAVEATS:
1. Due to recruitment difficulties, dosimetry data is limited.
2. Pre-clinical studies largely performed on porcine squamous esophageal epithelium as BE pre-clinical models are unavailable. Porcine esophageal wall layers are generally thinner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No